CLINICAL TRIAL: NCT06195735
Title: Forecasting Hypersensitivity Against PEG-asparaginase to Optimize Outcome in ALL
Status: Completed | Type: Observational
Sponsor: Aarhus University Hospital (Other)
Collaborators: Uppsala University (Other); University of Aarhus (Other)
Responsible Party: Principal Investigator, Birgitte Klug Albertsen, MD, PhD, Professor (Pediatric Hematology/Oncology), Aarhus University Hospital
Other Study IDs: Asp_pharmacokinetic-model
Record Dates: First submitted 2023-12-14; First posted 2024-01-08 (Actual); Last update posted 2024-01-08 (Actual); Status verified 2024-01

CONDITIONS: Acute Lymphoblastic Leukemia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 323 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Asparaginase is a cornerstone in the treatment of acute lymphoblastic leukemia (ALL). Clinical hypersensitivity reactions and PEG-asparaginase inactivation is common (12-13% of the patients on the NOPHO (Nordic Society for Paediatric Haematology and Oncology) ALL2008 protocol) and has become even more frequent after changing to the current Western European ALL Treatment protocol ALLTogether, despite the PEG coat, leading to increased asparaginase clearance and treatment truncation. Suboptimal anticancer therapy occurs in an additional 3-4% of the patients, who encounter expedited asparaginase clearance but no allergy symptoms (silent inactivation).

The aim of this study is to validate and potentially refine an already existing PEG-asparaginase pharmacokinetic model on data from patients treated according to the A2G main protocol.

DETAILED DESCRIPTION:
In comparison to the previous NOPHO ALL2008 protocol, the current A2G protocol aims at reducing the treatment intensity for patients with a good prognosis. More than 50% of the patients do no longer receive anthracyclines during induction therapy in order to avoid cardiotoxicity, and therefore the treatment relies more on PEG-asparaginase, which is given earlier than in previous NOPHO protocols. This underlines the additional importance of adequate asparaginase activity during the treatment period in order to have optimal treatment response on the predefined stratification days. Individual measurements (TDM) can help to identify patients with suboptimal activity and enable initiation of corrective measures, where current guidelines recommend an effective PEG-asparaginase trough concentration of ≥100 IU/L. In case of inactivation, patients are switched to the second line asparaginase formulation Erwinase, which is both expensive and very burdensome for the patients and hospitals because of need for frequent treatment. Patients that have their treatment truncated, have inferior outcome.

The present Western European ALL Treatment protocol ALLTogether (A2G) opened November 2018 as a pilot protocol in NOPHO, where 17% of the patients experienced hypersensitivity (14% clinical reactions and 3% silent inactivation). Early detection of allergic reactions and inactivity is important to avoid potential life threatening allergic reactions and a suboptimal treatment. Our study group has developed a PEG-asparaginase pharmacokinetic model to predict potential allergy and inactivation based on data from the A2G pilot protocol. Since then, the PEG-asparaginase treatment was changed due to inacceptable overall toxicity, which has now resulted in a doubling of hypersensitivity reactions. Hence, the pattern of enzyme clearance and immunogenicity may have changed.

Identification and prediction of increased clearance through asparaginase measurements during treatment will allow for early treatment adaptation, i.e., before suboptimal plasma levels have been reached. Timely identification of drug inactivation and treatment adaptation would therefore have potential to improve treatment outcome for a substantial number of the patients. The investigators aim to tackle this problem through pharmacokinetic-pharmacodynamic characterization of the relationships between dosage, asparaginase exposure and appearance of allergy symptoms in patients treated according to the A2G main protocol. This integrated knowledge can help facilitate development of tailored treatment strategies for individual patients.

ELIGIBILITY:
Inclusion Criteria:

* Treated for acute lymphoblastic leukemia (ALL) on the ALLTOGETHER main protocol

Exclusion Criteria:

* None

Max Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: All patients with ALL 1-45 years of age treated on the ALLTOGETHER main protocol in the Nordic and Baltic countries.
Sampling Method: Non-Probability Sample
Enrollment: 649 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
Number of participants with hypersensitivity Clinical allergy / silent inactivation | 2020-2023
  Patients with allergic reactions or silent inactivation

CONTACTS AND LOCATIONS:
Overall Officials: Birgitte K Albertsen, M.D., Principal Investigator — Aarhus University Hospital, Denmark
Locations (1):
- Aarhus University Hospital, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: No